CLINICAL TRIAL: NCT07010250
Title: Epithelial Dysmetabolism and Renal Fibrosis in ANCA Vasculitis
Acronym: PROTECT-Fi
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211383; PRTS-21-0009 (Other Grant/Funding Number: Ministry of health, France)
Record Dates: First submitted 2025-05-05; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: ANCA Associated Vasculitis; Extramembranous Glomerulopathy; Nephrotic Syndrome, Minimal Change; Interstitial Nephritis; IgA Nephropathy; Segmental Hyalinosis; Diabetic Nephropathies
Keywords: nephropathy; cohort
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Glomerulonephritis, Membranous; Nephrosis, Lipoid; Nephritis, Interstitial; Glomerulonephritis, IGA; Glomerulosclerosis, Focal Segmental; Diabetic Nephropathies; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Additional research analyzes on the care biopsy specimen, DNA, serum and plasma biobank, urine samples for lipidomic sudies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- ANCA Associated Vasculitis: Case
- Extramembranous Glomerulopathy: Control
- Nephrotic Syndrome, Minimal Change: Control
- Interstitial Nephritis: Control
- IgA Nephropathy: Control
- Segmental Hyalinosis: Control
- Diabetic Nephropathy: Control

SUMMARY:
The project is to explore in humans the hypothesis of the link between the alteration of tubulo-interstitial metabolism and the rate of deterioration of renal function by comparing various nephropathies.

DETAILED DESCRIPTION:
Patients with ANCA vasculitis with rapidly progressive glomerulonephritis with "crescent" will be compared to six other groups made up of patients with another nephropathy 1/extramembranous glomerulonephritis and 2/ nephropathy with minimal glomerular lesion (LGM) characterized by the absence of significant tubulointerstitial fibrosis lesions and slow evolution towards end-stage chronic renal failure ). Other groups of patients will 3/have interstitial nephropathy, 4/IgA mesangial glomerulopathy , 5/diabetic nephropathy, or 6/collapsing focal segmental hyalinosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for initial diagnostic PBR on native kidney
* 18 ans ≥ Age ≤ 90 ans
* Affiliation to french health insurance
* Patient having given consent

For the ANCA vasculitis group:

• Diagnosis of ANCA vasculitis retained on renal biopsy with ANCA anti-proteinase 3 (PR3) or ANCA anti-myeloperoxidase (MPO)

For the control groups:

• Diagnosis retained after the renal biopsy

* Interstitial Nephritis
* Or glomerular nephropathy such as minimal change nephropathy
* Or Segmental hyalinosis in itscollapsing form
* Or Extramembranous Glomerulopathy,
* Or glomerulopathy with mesangial IgA deposits
* Or diabetic nephropathy.

Exclusion Criteria:

* Kidney transplant patient
* Patient on dialysis (hemodialysis or peritoneal dialysis)
* Patient under legal protection, guardianship or curatorship
* Pregnancy or breastfeeding
* Enrollement in an interventional study except studies relating to ANCA vasculitis and nephropathy with mesangial IgA deposits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ANCA Associated Vasculitis The project is to test in humans the hypothesis of the link between the alteration of tubulo-interstitial metabolism and the rate of deterioration of renal function by comparing various nephropathies. A group of patients with ANCA vasculitis with rapidely progressive glomerulonephritis with "crescent" will be compared to six other groups : Patients with extramembranous Glomerulopathy and 2/ nephropathy with minimal glomerular lesion (LGM) by the absence of significant tubulointerstitial fibrosis lesions slow evolution towards end-stage chronic renal failure ). Other groups of patients will 3/have interstitial nephropathy, 4/IgA mesangial glomerulopathy , 5/diabetic nephropathy, or 6/collapsing focal segmental hyalinosis.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2029-06-02 (Estimated); Study Completion 2029-06-02 (Estimated)

PRIMARY OUTCOMES:
Spatial lipidomics for measuring tubular dysmetabolism | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured either through biospy at baseline or from blood and urine samples taken at baseline, after 15 days, 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  Their contribution for classifying ANCA vasculitis and other nephropathies will be evaluated.
Co-staining for measuring tubular segments markers | Through study completion up to end of study, when the last patients completed 1 year follow-up
  Measured either through biospy at baseline or from blood and urine samples taken at baseline, after 15 days, 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  Their contribution for classifying ANCA vasculitis and other nephropathies will be evaluated.
Immunofluorescence (at the protein level) for measuring peroxisome Proliferator-Activated Receptor-Gamma (PPAR-gamma) | Through study completion up to end of study, when the last patients completed 1 year follow-up
  Measured either through biospy at baseline or from blood and urine samples taken at baseline, after 15 days, 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  Its contribution for classifying ANCA vasculitis and other nephropathies will be evaluated.
Spatial transcriptomics (at the mRNA level) for measuring peroxisome Proliferator-Activated Receptor-Gamma (PPAR-gamma) | Through study completion up to end of study, when the last patients completed 1 year follow-up
  Measured either through biospy at baseline or from blood and urine samples taken at baseline, after 15 days, 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  Its contribution for classifying ANCA vasculitis and other nephropathies will be evaluated.

SECONDARY OUTCOMES:
Glomerular filtration rate evolution | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  CKDepi (Chronic Kidney Disease - EPIdemiology, a method for estimating glomerular filtration rate) decline.
  It is calculated with a patient's age, sexe and color of their skin as well as serum creatinine rates found in urine and blood samples.
  Measured at baseline, after 15 days, 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to study the differences of glomerular filtration rate evolution between patients with ANCA vasculitis and those with other nephropathies.
Urinary protein/creatinine ratio evolution | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured in urinary morning sample taken at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to :
  * group patients with similar characteristics in homogeneous groups.
  * study the differences in the evolution between patients with ANCA vasculitis and those with other nephropathies.
  * identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Urinary albumin/creatinine evolution ratio | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured in urinary morning sample taken at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to :
  * group patients with similar characteristics in homogeneous groups.
  * study the differences in the evolution between patients with ANCA vasculitis and those with other nephropathies.
  * identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Lipidomic analysis | Through study from baseline until one year visit.
  Measured in urinary morning sample taken at baseline, after 15 days, 2 months, 6 months and one year.
  More specifically there will be an anatomopathological analysis of lipid content (oil red o, Luxol blue, Nile red staining).
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Metabolomic analysis | Through study from baseline until one year visit.
  Measured in urinary morning sample taken at baseline, after 15 days, 2 months, 6 months and one year.
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Proportion of fibrotic tissues | At baseline.
  Measured in % with biopsy at the beginning of study. It will be used to study the impact of interstitial fibrosis in the relation between tubular dysmetabolism and ANCA vasculitis against other nephropathies.
Capillary density | At baseline.
  Measured with biopsy at the beginning of study. It will be used to study the impact of interstitial fibrosis in the relation between tubular dysmetabolism and ANCA vasculitis against other nephropathies
Markers of podocytes, renal epithelial cells and specific leukocyte populations | At baseline.
  Measured with biopsy at the beginning of study. It will be used to study the impact of interstitial fibrosis in the relation between tubular dysmetabolism and ANCA vasculitis against other nephropathies
Quantification of fibrosis | At baseline.
  Measured with biopsy at the beginning of the study, by Sirius Red staining. It will be used to study the impact of interstitial fibrosis in the relation between tubular dysmetabolism and ANCA vasculitis against other nephropathies
IMC (imaging mass cytometry) | At baseline.
  Tubular cell labeling with dedifferentiation at the beginning of study. It will be used to study the impact of interstitial fibrosis in the relation between tubular dysmetabolism and ANCA vasculitis against other nephropathies.
Transcriptomic analysis | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured with biopsy at the beginning of study and blood sample taken at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  More specifically an anatomopathological analysis with single cell transcriptomic analyses along a study of gene expression (epigenetic deregulation) will be carried out.
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Diastole | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured in mmHg (average of 3 measures) at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Systole | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured in mmHg (average of 3 measures) at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Heart rate | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured in beat per minute (average of 3 measures) at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Blood count analysis | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measures on leukocytes, red blood cells and platelets with blood samples taken at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  It will be used to group patients with similar characteristics in homogeneous groups and identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
Leukocytes evolution | Through study completion up to end of study, when the last patients completed 1 year follow-up.
  Measured in several ways :
  * by blood count with blood samples taken at baseline, after 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up
  * through anatomopathological analysis by IMC with the biopsy core taken at the beginning of the study
  * specific leukocytes population will be studied for interstitial fibrosis assessment Measured at baseline, after 15 days, 2 months, 6 months and then every 6 months until the last patients completed 1 year follow-up.
  They will be used to :
  * study the differences in the evolution between patients with ANCA vasculitis and those with other nephropathies.
  * identify similaritites in patients trajectories according to which nephropathy they were diagnosed with.
  * study the impact of interstitial fibrosis in the relation between tubular dysmetabolism and ANCA vasculitis against other nephropathies.

CONTACTS AND LOCATIONS:
Overall Officials: Marine LIVROZET, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Georges-Pompidou European Hospital, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).